CLINICAL TRIAL: NCT01885975
Title: Personality Profile of Patients With Apical Ballooning Syndrome (ABS)
Brief Title: Personality Profile of Patients With Apical Ballooning Syndrome
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Abhiram Prasad, PI, Mayo Clinic
Other Study IDs: 13-003419
Record Dates: First submitted 2013-06-20; First posted 2013-06-25 (Estimated); Last update posted 2015-02-16 (Estimated); Status verified 2015-02

CONDITIONS: Apical Ballooning Syndrome
Keywords: Apical Ballooning syndrome; Personality
MeSH Terms: conditions — Takotsubo Cardiomyopathy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators' hypothesis is that patients with apical ballooning syndrome (ABS) will manifest a personality profile that differs than that of a population of similar range of ethnic and socioeconomic status.

ELIGIBILITY:
Inclusion criteria:

1. Patients who have suffered with ABS
2. Adults (18 years or older)
3. Able to read English at a 6th grade level (questionnaires are self-administered and written in English)

Exclusion criteria:

1. Have withdrawn from the registry
2. Have died

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will be conducted among participants in the Mayo Clinic Apical Ballooning Registry. These patients were prospectively diagnosed with Apical Ballooning Syndrome at the time of presentation with their acute illness, and consented to participation in a registry. They are residents of Olmsted County, and the surrounding regions for which the Mayo Clinic serves as a tertiary care center. Enrollment in the registry requires satisfaction of standard criteria for the diagnosis of ABS and includes the administration of a standardized questionnaire. Subjects have agreed to participate in yearly follow up questionnaires about their health status.
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2013-07; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Range of personality traits as assessed by the "NEO-PI-3" | Baseline: the traits will be assessed once upon enrollment into the study
  The "NEO PI-3" measures the five major domains of personality, which are:
  * Neuroticism
  * Extraversion
  * Openness
  * Agreeableness
  * Conscientiousness

CONTACTS AND LOCATIONS:
Overall Officials: Abhiram Prasad, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States